CLINICAL TRIAL: NCT06054347
Title: Standardized Evaluation of Long-term Neurocognitive Development of Children From Age 3 With Pyridoxine Dependent Epilepsy by Antiquitine Deficiency
Brief Title: Evaluation by a Vineland II Scale of Long-term Development of Children With Pyridoxine Dependent Epilepsy
Acronym: EPIDEV-B6
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC23_0181
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Pyridoxine-Dependent Epilepsy
MeSH Terms: conditions — Pyridoxine-dependent epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: VINELAND II — Standardised questionnaire filled by the investigator during an interview with the parents or with the patient himself if capable of it. Duration 1 hour to 1 hour and a half.

SUMMARY:
This study aims to evaluate with the VINELAND II scale the long-term neurocognitive development of children above age 3 years with pyridoxine dependent epilepsy related to antiquitine deficiency.

DETAILED DESCRIPTION:
Pyridoxine dependent epilepsy related to antiquitine deficiency is a rare and severe genetic epilepsy that usually starts within the first month of life. The treatment is based on high dose of Vitamin B6 (Pyridoxine) which is usually highly effective to control the seizures. However, most patients show impaired neurodevelopment.

Ten years ago, international recommendations have changed and a lysine restricted diet was added as an adjunct therapy with the hope to improve neurodevelopment.

Very few studies have evaluated the cognitive development of these patients in a standardized way, and these studies evaluate very few patients.

It seems therefore essential to study in a standardized way the neurocognitive development of these patients in order to evaluate the impact of the care.

The VINELAND adaptative behaviour scale II has been chosen because it can evaluate a patient whatever the age or the intellectual abilities through a semi-structured questionnaire completed with the parents, and gives a wide view of the neurocognitive development and everyday life autonomy of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age above 3 years old
* Pyridoxine dependent epilepsy genetic diagnosis (mutation in ALDH7A1 gene)
* No objection of the patient or his legal representatives.

Exclusion Criteria:

* Poor understanding of French language.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of patients diagnosed with pyridoxine dependent epilepsy and already published (Gibaud et al) completed with new cases.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Vineland II Adaptive Behaviour scales (VABS) total mean score and subscale mean scores | Baseline
  Standardized questionnaire filled by the investigator during an interview with the parents or the patient himself if possible. 5 domains. Maximum score 160, minimum score 20, mean score 100, standard deviation 15

SECONDARY OUTCOMES:
Determine if the treatments actually used for patients with pyridoxine dependent epilepsy have an impact on their long-term neurocognitive development, especially the lysine restricted diet | Baseline
  Questionnaire filled by the investigator during an interview with the parents or the patient himself if possible
Evaluation of executive functions with the BRIEF scale | Baseline
  Questionnaire filled by the investigator during an interview with the parents or the patient himself if possible. 87 questions. 15 minutes duration.
Clinical and para-clinical description of the population studied | Baseline
  Questionnaire filled by the investigator during an interview with the parents or the patient himself if possible.
genotype phenotype correlation | baseline
  study the genotype phenotype correlation in the light of patient long term neurocognitive development

CONTACTS AND LOCATIONS:
Overall Officials: Patrick VAN BOGAERT, PhD - MD, Principal Investigator — University Hospital, Angers
Locations (12):
- France (12):
  - CHU Angers, Angers
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - CHRU Morvan, Brest
  - CHU d'Estaing, Clermont-Ferrand
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital de la Timone-Enfants, Marseille
  - CHU Gui de Chautiac, Montpeliier
  - Hôpital Necker-Enfants malades, Paris
  - Centre Hospitalier Saint Nazaire, Saint-Nazaire
  - CHU Toulouse, Toulouse
  - Hôpital Clocheville, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coughlin CR 2nd, Swanson MA, Spector E, Meeks NJL, Kronquist KE, Aslamy M, Wempe MF, van Karnebeek CDM, Gospe SM Jr, Aziz VG, Tsai BP, Gao H, Nagy PL, Hyland K, van Dooren SJM, Salomons GS, Van Hove JLK. The genotypic spectrum of ALDH7A1 mutations resulting in pyridoxine dependent epilepsy: A common epileptic encephalopathy. J Inherit Metab Dis. 2019 Mar;42(2):353-361. doi: 10.1002/jimd.12045. Epub 2019 Feb 22. PMID 30043187
- [Background] Wilson MP, Plecko B, Mills PB, Clayton PT. Disorders affecting vitamin B6 metabolism. J Inherit Metab Dis. 2019 Jul;42(4):629-646. doi: 10.1002/jimd.12060. Epub 2019 Mar 20. PMID 30671974
- [Background] Basura GJ, Hagland SP, Wiltse AM, Gospe SM Jr. Clinical features and the management of pyridoxine-dependent and pyridoxine-responsive seizures: review of 63 North American cases submitted to a patient registry. Eur J Pediatr. 2009 Jun;168(6):697-704. doi: 10.1007/s00431-008-0823-x. Epub 2008 Sep 2. PMID 18762976
- [Background] Baxter P. Epidemiology of pyridoxine dependent and pyridoxine responsive seizures in the UK. Arch Dis Child. 1999 Nov;81(5):431-3. doi: 10.1136/adc.81.5.431. PMID 10519720
- [Background] Coughlin CR 2nd, Tseng LA, Abdenur JE, Ashmore C, Boemer F, Bok LA, Boyer M, Buhas D, Clayton PT, Das A, Dekker H, Evangeliou A, Feillet F, Footitt EJ, Gospe SM Jr, Hartmann H, Kara M, Kristensen E, Lee J, Lilje R, Longo N, Lunsing RJ, Mills P, Papadopoulou MT, Pearl PL, Piazzon F, Plecko B, Saini AG, Santra S, Sjarif DR, Stockler-Ipsiroglu S, Striano P, Van Hove JLK, Verhoeven-Duif NM, Wijburg FA, Zuberi SM, van Karnebeek CDM. Consensus guidelines for the diagnosis and management of pyridoxine-dependent epilepsy due to alpha-aminoadipic semialdehyde dehydrogenase deficiency. J Inherit Metab Dis. 2021 Jan;44(1):178-192. doi: 10.1002/jimd.12332. Epub 2020 Dec 1. PMID 33200442
- [Background] Tourrette C., Evaluer les enfants avec déficiences ou troubles du développement. PARIS : Dunod, 2006
- [Background] Fombonne E. ; Achard S. ; Tuffreau R. L'évaluation du comportement adaptatif : l'échelle de Vineland. In Handicap et inadaptations. Les Cahiers du CTNERHI, n° 67-68, juil. / déc. 1995. p. 79-90.3
- [Background] Gioia GA, Isquith PK, Guy SC, Kenworthy L. The Behaviour Rating Inventory of Executive Function. Lutz, FL: Psychological Assessment Resources; 2000.
- [Background] Gibaud M, Barth M, Lefranc J, Mention K, Villeneuve N, Schiff M, Maurey H, Barthez MA, Caubel I, Chouchane M, Doummar D, Kossorotoff M, Lamblin MD, Roubertie A, Nabbout R, Van Bogaert P. West Syndrome Is an Exceptional Presentation of Pyridoxine- and Pyridoxal Phosphate-Dependent Epilepsy: Data From a French Cohort and Review of the Literature. Front Pediatr. 2021 Mar 5;9:621200. doi: 10.3389/fped.2021.621200. eCollection 2021. PMID 33748042